CLINICAL TRIAL: NCT01471613
Title: Safety and Effect of Lithium, Umbilical Cord Blood Cells and the Combination in the Treatment of Acute and Sub-acute Spinal Cord Injury : a Randomized, Double-Blinded Placebo-Controlled Clinical Trial
Brief Title: Lithium, Cord Blood Cells and the Combination in the Treatment of Acute & Sub-acute Spinal Cord Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: China Spinal Cord Injury Network (Network)
Collaborators: Chengdu PLA General Hospital (Other); StemCyte, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN102c
Record Dates: First submitted 2011-10-12; First posted 2011-11-15 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; umbilical cord blood cell; cell transplant; lithium carbonate
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Lithium Carbonate; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Group C - Cord blood cell (Experimental): Conventional treatment, cord blood cell transplant and placebo
  Interventions: Procedure: Conventional Treatment; Biological: Cord Blood Cell; Other: Placebo
- Group A - Control (Placebo Comparator): Conventional treatment and placebo
  Interventions: Procedure: Conventional Treatment; Other: Placebo
- Group B - Lithium Carbonate (Experimental): Conventional treatment and lithium carbonate
  Interventions: Procedure: Conventional Treatment; Drug: Lithium Carbonate Tablet
- Group D - Combination Therapy (Experimental): Conventional treatment, cell transplant and 6-weeks course of lithium carbonate
  Interventions: Procedure: Conventional Treatment; Drug: Lithium Carbonate Tablet; Biological: Cord Blood Cell

INTERVENTIONS:
Procedure: Conventional Treatment — Conventional treatment includes surgeries such as laminectomy, spinal decompression etc. and the medicine generally adapted to treat spinal cord injury
Drug: Lithium Carbonate Tablet — 250mg/tablet, administrated orally for 6 weeks.
  Arms: Group B - Lithium Carbonate; Group D - Combination Therapy
Biological: Cord Blood Cell — Cord blood mononuclear cell, 6.4 million viable cells, are transplanted into spinal cord at upper and lower edges of the injured site
  Arms: Group C - Cord blood cell; Group D - Combination Therapy
Other: Placebo — Placebo tablet, orally administration of placebo for 6 weeks
  Arms: Group A - Control; Group C - Cord blood cell

SUMMARY:
The trial is to investigate the safety and efficacy of oral lithium, intraspinal umbilical cord blood mononuclear cell transplant, and the combination in the treatment of acute and subacute spinal cord injury

ELIGIBILITY:
Inclusion Criteria:

* either gender and 18-65 years old;
* acute or subacute traumatic spinal cord injury (defined as SCI resulting from an exteneral non-penetrating cause that occurred within 4 weeks);
* neurological status of ASIA A;
* neurological level between C5-T11;
* MRI shows injury site is within 3 vertebral level and necrotic focus, if exist, is less than 1/3 of the spinal cord diameter;
* professional judgment determinate that subjects need a spinal decompression surgery;
* subjects able to complete neurological examination;
* subjects have voluntarily signed and dated an informed consent form.

Exclusion Criteria:

* penetration SCI such as gun-shoot, knife-cutting or SCI caused by non-traumatic conditions;
* spinal cord lesion exceeds three segments or necrotic focus with diameter larger than 1/3 of the spinal cord;
* severe complications;
* significant medical diseases or infection;
* pregnant or lactating woman, or female of childbearing potential and who is unwilling to use an effective contraceptive method while enrolled in the study;
* unavailability of suitable umbilical cord blood cells;
* contraindication of lithium carbonate and/or spinal decompression surgery
* subject is currently participating in another study or has been taking any investigational drug within the last 4 weeks prior to screening;
* investigator suggests that the subject would not be suitable to participate this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in AIS Motor and sensory scores and ASIA Impairment Scales in 48 weeks | Week 0, 1, 2, 6, 14, 24 and 48

SECONDARY OUTCOMES:
Walking | Week 2, 6, 14, 24, 48
  Walking Index of Spinal Cord Injury (WISCI)
Functional assessment | Week 2, 6, 14, 24, 48
  Spinal Cord Injury Measure (SCIM) Score
Locomotion | Week 2, 6, 14, 24, 48
  Kunming locomotor scales
Spasticity grade | Week 2, 6, 14, 24, 48
  Modified Ashworth Scale
Pain | Week 2, 6, 14, 24, 48
  Numerical rating scales

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhu, MD, Principal Investigator — Chengdu PLA General Hospital
Locations (1):
- Treating Center of Spinal Cord Injury, Chinese PLA Chengdu Army Kunming General Hospital, Kunming, Yunnan, China